CLINICAL TRIAL: NCT05990543
Title: Combination of Nelmastobart and Capecitabine Therapy in Metastatic Colorectal Cancer With Resistance or Intolerance to Oxaliplatin and Irinotecan-based Chemotherapy - A Single Arm, Phase 1b/2, Multicenter Study
Brief Title: Combination of Nelmastobart and Capecitabine Therapy in Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Lee, Soo Hyeon, Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NelCap001
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Recurrent or Metastatic Colorectal Cancer
Keywords: colorectal cancer; immunotherapy
MeSH Terms: conditions — Recurrence; Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Nelmastobart + Capecitabine
  Interventions: Drug: Nelmastobart and Capecitabine

INTERVENTIONS:
Drug: Nelmastobart and Capecitabine — Nelmastobart intravenously every 3 weeks until PD or discontinuation due to toxicity. Administered on Day 1 of each cycle.
  Capecitabine is administered orally for two weeks followed by a one-week rest period

SUMMARY:
This is an open-label clinical trial aimed at evaluating the safety and efficacy of the combination treatment of nelmastobart with capecitabine in patients diagnosed with metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is the third most commonly diagnosed cancer in men and the second most common cancer in women worldwide, with an estimated 1.9 million new cases and 935,000 deaths in 2020, according to the World Health Organization. Patients with metastatic colorectal cancer typically undergo first-line treatment consisting of fluorouracil-based chemotherapy (oxaliplatin and irinotecan) with or without vascular endothelial growth factor (VEGF)-based therapy (primarily bevacizumab), and epidermal growth factor receptor (EGFR)-targeted therapies (in patients with RAS wild-type tumors). Second-line treatment options may include alternative chemotherapy regimens. Third-line treatment options are often limited for patients with metastatic colorectal cancer, as they tend to exhibit poor objective response rates and short progression-free survival. However, despite their good performance status, patients often encounter limited options for third-line treatment, resulting in a daunting and frustrating situation.

This study will enroll patients aged ≥18 years who are resistant or intolerant to oxaliplatin and irinotecan-based chemotherapy. The study will evaluate the safety of the Nelmastobart and capecitabine combination therapy in Phase 1b. After identifying the Recommended Phase 2 Dose (RP2D), the study will assess the efficacy of the Nelmastobart and capecitabine combination therapy in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥18 years of age at the time of signing the informed consent form (ICF).
2. Subjects with histologically or cytologically confirmed colorectal adenocarcinoma who have failed or are ineligible for oxaliplatin and irinotecan-based chemotherapy.
3. Subjects with advanced/metastatic solid tumors, with evaluable lesion as determined by Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.

   Measurable lesion is optional.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤2.
5. Adequate organ and bone marrow function characterized by the following at screening:

   1. Absolute neutrophil count(ANC) ≥1.0 × 109/L;b.
   2. Platelets ≥75 × 109/L;c.
   3. Hemoglobin ≥9.0 g/dL (with or without blood transfusions).
   4. Adequate renal function defined by Serum creatinine ≤ ULN x 1.5 or an estimated creatinine clearance ≥30 mL/min according to the Cockcroft Gault formula or by 24-hour urine collection for creatinine clearance, or according to local institutional standard method.
   5. Serum total bilirubin ≤2.0 x upper limit normal (ULN), if a subject with biliary obstruction is considered suitable if they meet the criteria after appropriate bile drainage.
   6. ALT and AST ≤ 3 × ULN, or ≤5 × ULN in the presence of liver metastases.
6. Adequate cardiac function: QTc ≤480 msec; if QTc exceeds 480 msec, subjects can be enrolled if the average QTc value is less than 480 msec by measuring 3 times consecutively in total.
7. The subject is able to swallow and retain oral medication
8. Serum β hCG test negative within 14 days before the first administration of the study treatment (women of childbearing potential only)
9. Requirement for contraception must be observed by the subject.

   * Eligible women (all women of reproductive potential who are either undergoing clinical trial treatment or within 4 weeks after discontinuing clinical trial treatment, and who are not using appropriate contraception) must use the following contraceptive methods to be eligible for enrollment.
   * Subjects must abstain from all forms of sexual intercourse and are encouraged to practice consistent abstinence in their daily lives. Periodic abstinence methods (e.g., calendar-based methods, cervical mucus observation, basal body temperature methods, etc.) and withdrawal are not considered acceptable contraceptive methods.
   * Accepted infertility surgical procedures: Bilateral oophorectomy with or without hysterectomy; Tubal ligation at least 6 weeks before enrollment in this clinical trial. Bilateral oophorectomy is only allowed if the subject's potential for pregnancy is confirmed through hormone level assessment.
   * In the case of female participants in the clinical trial, their male partners who have undergone vasectomy (screening performed at least 6 months prior) should be their exclusive partners during the participation in this clinical trial
   * During the clinical trial, male participants should use condoms during sexual intercourse while they are receiving the investigational drug and for up to 1 month after discontinuing the treatment (after the last dose).
10. Life expectancy of at least 12 weeks. Capable and willing to give signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
11. Subject has signed the Informed Consent Form (ICF) prior to any screening procedures being performed

Exclusion Criteria:

1. Patient has a known or suspicious hypersensitivity to fluoropyrimidines.
2. Any cytotoxic chemotherapy from a previous treatment regimen within 14 days. If the subject received an investigational drug from another clinical trial, the subject can be enrolled after 2 weeks of last administration and more than 5 x half-life of the investigational drug. If monoclonal antibody therapy was given, the subject can be enrolled after four weeks after the last dose.
3. Uncontrolled severe infection
4. Subjects with conditions requiring high doses of steroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive medications are excluded, all of the following will not be excluded:

   1. Brief (<7 days) use of systemic corticosteroids is allowed when use is considered standard of care.
   2. Subjects requiring intermittent use of bronchodilators, inhaled steroids, or local steroid injections will not be excluded.
   3. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
5. Subjects who are pregnant or breastfeeding women.
6. History of autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Subjects with vitiligo, psoriasis not requiring systemic treatment, type 1 diabetes mellitus, hypothyroidism stable with hormone replacement, Sjögren's syndrome, or resolved childhood asthma/atopy will not be excluded.
7. Active central nervous system (CNS) lesions (i.e., those with radiologically unstable or symptomatic brain lesions). For those who receive radiation or surgical treatment, the subject can be enrolled if the subject is maintained without steroid therapy and the evidence of CNS disease progression for more than 4 weeks. However, patients with leptomeningeal metastases are excluded.
8. Subjects with a documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class IV within 6 months prior to screening.
9. Subjects with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan.
10. Subjects who have received a prior allogeneic stem cell or solid organ transplant.
11. Subjects who have received a live attenuated vaccine within 30 days prior to screening. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
12. History of other primary cancer. Exceptions are as follows:

    - Adequately treated non-melanoma skin cancer (basal cell or squamous cell carcinoma), curatively treated in situ cancer of the cervix or stage I bladder cancer, completely resected thyroid cancer without distant metastasis in which all treatment has been completed (Appropriate wound healing is required prior to clinical trial enrollment)
13. Subject has not recovered to ≤ grade 1 (except alopecia) from related adverse effects of any prior anticancer therapy.
14. Radiotherapy with a wide field (more than 30% of the bone marrow) of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment.
15. Subject who has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from adverse effects of such procedure.
16. Subjects with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of capecitabine.
17. Subjects who have known active hepatitis B (defined as positive hepatitis B surface antigen [HBsAg] with detected hepatitis B virus [HBV] DNA) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
18. Subjects with genetic conditions such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
19. As judged by the Investigator, all other symptoms and associated disease for which the investigator determined that participation in this study is contraindicated (e.g. Infection/inflammation; severe liver dysfunction; bilateral diffuse interstitial lung disease; uncontrolled renal disease; unstable heart and lung disease; hemorrhagic disease; intestinal obstruction; unable to swallow oral pills; social and psychological problems, etc.)
20. Medical, psychiatric, cognitive, or other conditions that may interfere with the ability of the subject to understand the subject information, provide the informed consent, follow the protocol process, or complete the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to approximately 2 years
  The MTD was defined as the highest dose at which no dose limiting toxicity (DLT) was experienced by the first 3 patients in that cohort, or the dose at which a DLT was experienced by no more than 1 of 6 patients evaluable for toxicity.
Progression free survival | Up to approximately 2 years
  PFS events is defined as the interval from the first dose of investigational treatment to the earlier of the first documentation of objective progressive disease (PD) or death from any cause,whichever comes first.

SECONDARY OUTCOMES:
Overall response rate | Up to approximately 2 years
  ORR is defined as the proportion of participants who achieve a CR or PR as assessed by RECIST v1.1.
Overall survival | Up to approximately 2 years
  Progression free survival (PFS) will be calculated from the first dose of investigational treatment until date of progression or death without progression, using the Kaplan-Meier method accompanied by determination of the median and its 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Medical Center 73, Goryeodae-ro, Seongbuk-gu, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No